CLINICAL TRIAL: NCT03247179
Title: Secondary Prevention With the Mobile PTSD Coach App to Improve Health Outcomes and the Continuity of Care Following Traumatic Physical Injury: A Randomized Controlled Trial
Brief Title: The Mobile PTSD Coach App in Acute Injury Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Maria Pacella, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO16010595
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain; Acute Pain Due to Trauma; Posttraumatic Stress Disorder
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental condition (PTSD Coach app usage), or the treatment as usual condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD Coach Condition (Experimental): PTSD Coach App
  Interventions: Other: PTSD Coach mobile application
- Treatment as Usual Condition (No Intervention): Treatment as Usual

INTERVENTIONS:
Other: PTSD Coach mobile application — The PTSD Coach app is publicly available for free, and draws on cognitive behavioral therapy components to help participants learn, manage, and cope with their PTSD symptoms in real time.
  Arms: PTSD Coach Condition

SUMMARY:
This project is a preliminary randomized controlled trial testing the potential impact of the PTSD Coach mobile application at reducing posttraumatic stress and pain symptoms among acutely injured trauma patients. Immediately following the injury, patients will be randomly assigned to use the PTSD Coach app, or to the treatment as usual condition.

DETAILED DESCRIPTION:
Traumatic injury is the leading cause of mortality in the U.S. for young people, and a source of long-term morbidity in all ages. A majority of trauma patients report chronic pain (CP) and disability at 4-months (30%- 79%) and 12-months (63%) post-injury. Maladaptive psychological processes have a stronger association with the transition to CP than does injury severity. Posttraumatic stress disorder (PTSD) symptoms (e.g., intrusions, avoidance and hyperarousal) occur in up to 22% of post-injury patients and herald the transition from acute to CP. Although psychological interventions can modify PTSD symptoms, and reduce CP, it is unknown if early intervention to prevent PTSD symptoms can prevent post-injury CP altogether. "PTSD Coach" is a publicly available, free, mobile app that provides scalable and psychosocial support modeled on principles of cognitive-behavioral therapy. PTSD Coach has helped Veterans and civilians to manage PTSD.

This project will test whether PTSD Coach can reduce post-injury maladaptive psychological processes and thereby prevent post-injury CP. The preventive intervention will be targeted towards those at the highest-risk of developing PTSD.

The investigators propose to test the efficacy of the PTSD Coach app vs. treatment as usual (TAU) among a sample of acute physical injury patients, to: 1) Determine engagement with PTSD Coach, by measuring frequency of use over 4-weeks and assessing ratings of usefulness and qualitative feedback: it is expected that >80% of PTSD Coach users will use the app at least once a week, and will rate it as at least somewhat helpful; 2) Estimate effect on CP symptoms by measuring PTSD and pain intensity at 1- and 3-months. The effect of the intervention on pain interference, disability, and coping self-efficacy will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults seeking treatment in the ED
* Adults between the ages of 18-65
* Sustained a musculoskeletal injury (e.g., fractures, sprains or strains, contusions, dislocations, crushing injuries and open wounds; and other chief complains involving the neck, back, or extremities)
* Injury resulting from a motor vehicle crash (MVC) or motorcycle crash (MCC) that occurred within the past 24 hours
* Eligible patients must own a mobile phone with short-message service (SMS) features (e.g., the ability to send and respond to text messages) and the ability to download apps
* Participants must self-report that they experienced a potential traumatic event reflected by Criterion A of the DSM-5 PTSD diagnosis (endorse actual or perceived life threat and/or serious injury141,142)
* Participants must self-report that they experienced a painful injury reflected by a pain score ≥4 using the verbal numerical score (0-10) in response to the question: "On a scale of 0-10, how severe is your pain?"
* Patients with a past history of PTSD, but not currently receiving treatment (e.g., benzodiazepines or mental/behavioral therapy), are eligible for participation.

Exclusion Criteria:

* Presenting to the ED for a non-MVC/MCC (i.e., fall, assault)
* Participants who do not own a mobile phone with SMS features
* Participants with a pain score < 4 or do not endorse Criterion A of the DSM-5 PTSD diagnosis
* Spinal injuries
* Major lacerations resulting in significant damage to subcutaneous tissue (e.g., degloving) and specific nerve injury (these injuries could lead to a distinct neuropathic pain syndrome)
* Traumatic brain injury; Evidence of moderate to severe cognitive impairment secondary to trauma-related head injury (GCS<13)
* Self-inflicted injury
* Time since trauma > 24 hours
* Non-English speaking; younger than 18 or older than 65
* Not medically stable or alert and oriented
* Initiation of benzodiazepines and other psychotropic medications at time of ED visit
* Initiation of mental or behavioral health therapy at time of ED visit
* Currently enrolled in treatment (medication or mental/behavioral health therapy) for PTSD
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM 5 (Diagnostic and Statistical Manual for Mental Disorders-5) | past 30-days
  PTSD symptoms

SECONDARY OUTCOMES:
Short Form of the Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale | 7-days
  8-items assessing pain interference
Short Form of the PROMIS Pain Intensity Scale | 7-days
  3-items assessing pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Pacella, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan in place yet because it is undecided whether the research team will need to share the data with investigators/researchers not listed on the protocol.

REFERENCES:
- [Derived] Pacella-LaBarbara ML, Plaitano EG, Suffoletto BP, Kuhn E, Germain A, Jaramillo S, Repine M, Callaway CW. A longitudinal assessment of posttraumatic stress symptoms and pain catastrophizing after injury. Rehabil Psychol. 2023 Feb;68(1):32-42. doi: 10.1037/rep0000481. PMID 36821344
- [Derived] Brienza A, Suffoletto BP, Kuhn E, Germain A, Jaramillo S, Repine M, Callaway CW, Pacella-LaBarbara ML. The role of specific sources of social support on postinjury psychological symptoms. Rehabil Psychol. 2021 Nov;66(4):600-610. doi: 10.1037/rep0000388. Epub 2021 Aug 16. PMID 34398631
- [Derived] Pacella-LaBarbara ML, Suffoletto BP, Kuhn E, Germain A, Jaramillo S, Repine M, Callaway CW. A Pilot Randomized Controlled Trial of the PTSD Coach App Following Motor Vehicle Crash-related Injury. Acad Emerg Med. 2020 Nov;27(11):1126-1139. doi: 10.1111/acem.14000. Epub 2020 May 19. PMID 32339359